CLINICAL TRIAL: NCT00054873
Title: Tezacitabine With or Without 5-Fluorouracil (5-FU) for Advanced Esophageal Cancer or Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiron Corporation (Industry)
Purpose: Treatment
Other Study IDs: TEZ001
Record Dates: First submitted 2003-02-12; First posted 2003-02-13 (Estimated); Last update posted 2006-07-11 (Estimated); Status verified 2006-06

CONDITIONS: Esophageal Neoplasms; Stomach Neoplasms; Adenocarcinoma
Keywords: Adenocarcinoma of the esophagus or stomach
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Adenocarcinoma; Adenocarcinoma Of Esophagus | interventions — tezacitabine; Fluorouracil

INTERVENTIONS:
Drug: tezacitabine
Drug: 5-fluorouracil

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of tezacitabine when given alone or in combination with 5-fluorouracil (5-FU) to subjects who have advanced esophageal or gastric adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Males and females greater than or equal to 18 years of age.
* Histologically confirmed recurrent (inoperable) or metastatic adenocarcinoma of the esophagus, gastroesophageal junction, or stomach.
* At least one bidimensionally measurable lesion, not previously irradiated, with a diameter that meets RECIST criteria, that can be serially measured. Intraluminal tumors, evaluable only by endoscopy, are not acceptable as target lesions.
* Karnofsky Performance Score greater than or equal to 70%.
* Subjects must be in the second line therapy setting, thus they must have experienced progression following treatment with one (and only one) prior chemotherapy regimen used for the treatment of unresectable locally advanced, recurrent, or metastatic disease.
* Recovery from any serious (grade 3 or higher) toxic effects of prior radiation therapy.
* Adequate hematologic profile: absolute neutrophil count greater than or equal to 1,500/mm3; hemoglobin greater than or equal to 9 g/dL; hematocrit greater than or equal to 30% (transfusion allowed); and platelet count greater than or equal to 100,000/mm3.
* Adequate hepatic function: bilirubin less than or equal to 1.5 mg/dL; AST and ALT less that 2.5 X ULN (5 X ULN if liver involved with tumor); alkaline phosphatase less than 5 X ULN
* Adequate renal function; serum creatinine less than or equal to 1.5 mg/dL or calculated creatinine clearance greater than 50 mL/min.
* Both male and female subjects of childbearing potential must be using a contraceptive method that is medically acceptable to the investigative center.
* Disease-free from a prior malignancy, other than non-melanoma skin cancer or carcinoma in-situ of the cervix, for greater than 5 years.

Exclusion Criteria:

* Unstable angina or class III or IV New York Heart Association heart disease.
* CNS metastases.
* Pregnant or breast-feeding.
* Uncontrolled seizure disorder.
* Ongoing (grade 3 or higher) stomatitis, esophagopharyngitis, or uncontrolled diarrhea.
* Impaired nutritional status as evidenced by a serum albumin of 2.7 mg/dL or less.
* Major surgery, chemotherapy, immunotherapy, or radiotherapy during the 28 days preceding the first study treatment. Concomitant anticancer therapy (chemotherapy, immunotherapy, or radiation) or other investigational agents during study participation or 28 days prior to study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-11; Study Completion 2004-12

CONTACTS AND LOCATIONS:
Locations (29):
- United States (29):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - ACRC/Arizona Clinical Research Center, Tucson, Arizona
  - Glendale Memorial Hospital, Glendale, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Tower Hematology Oncology Medical Group, Los Angeles, California
  - Comprehensive Cancer Center at DRMC, Palm Springs, California
  - Desert Regional Medical Center, Palm Springs, California
  - Sharp Clinical Oncology Research, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Cancer Institute Medical Group, Santa Monica, California
  - Denver VAMC, Denver, Colorado
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Memorial Regional Comprehensive Cancer Center, Weston, Florida
  - Northwestern University, Feinberg School of Medicine, Division of Hematology/Oncology, Chicago, Illinois
  - The University of Chicago, Chicago, Illinois
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - LSU Health Sciences Center, Dept. of Medicine, Hematology/Oncology, Shreveport, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Josephine Ford Cancer Center, Henry Ford Health System, Detroit, Michigan
  - Kansas City Oncology and Hematology Group, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - The Sarah Cannon Cancer Center, Tennessee Oncology, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - University of Texas, MD Anderson Cancer Center, Houston, Texas
  - Swedish Cancer Institute, Seattle, Washington